CLINICAL TRIAL: NCT01730417
Title: Phase I Study of the Safety, Distribution, and Radiation Dosimetry of Ultratrace Iobenguane 123I-mIBG-Nanodosing: the Path to Higher Sensitivity and Lower Toxicity Radiopharmaceuticals
Brief Title: Phase I Study of the Safety, Distribution, and Radiation Dosimetry of Ultratrace Iobenguane 123I-mIBG
Acronym: mIBG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bennett Chin (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Molecular Insights Pharmaceuticals (Unknown)
Responsible Party: Sponsor-Investigator, Bennett Chin, Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00019124 (MIP-CA130394-01); 5R44CA130394-03 (NIH)
Record Dates: First submitted 2012-11-07; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Neuroendocrine Tumors; Heart Failure
Keywords: Phase 1; no carrier added metaiodobenzylguanidine; radiation dosimetry
MeSH Terms: conditions — Neuroendocrine Tumors; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation dosimetry (Experimental): no carrier added metaiodobenzylguanidine
  Interventions: Drug: no carrier added metaiodobenzylguanidine

INTERVENTIONS:
Drug: no carrier added metaiodobenzylguanidine — Sequential imaging was performed to determine radiation dosimetry of high specific activity 123I-mIBG
  Other Names: Ultratrace

SUMMARY:
The goal of this proposal is to produce and test high specific activity Ultratrace iobenguane I 123 in normal human volunteers.

DETAILED DESCRIPTION:
The goal of this proposal is to produce and test high specific activity Ultratrace iobenguane I 123 in normal human volunteers. The low specific activity iobenguane I 123 has been shown to be useful for the detection and staging of neuroendocrine tumors in adults and children and imaging neuronal activity in the heart. The innovation in this proposal is through the use of patented solid phase technology to produce a proven diagnostic agent at extremely high specific activity to increase sensitivity and specificity and lower radiation exposure to normal organs without the pharmacologically active cold carrier compound. The FDA considers iobenguane labeled with two different isotopes of iodine [I-131 and I-123] as two distinct drugs requiring distinct regulatory applications.

To meet the required quality standards for the chemistry, manufacturing and controls component of an IND application, GMP quality polymer drug precursor is used to generate the Ultratrace diagnostic iodine-123 agent. Analytical methods were validated with the proposed final drug formulation to demonstrate the final drug does not interfere with tests used to define the identity, purity, and strength of the agent. The drug product was verified for apyrogenicity and sterility before human testing. The IND application was written and submitted to the FDA and the Duke Medical Center IRB. MIP produces clinical trial material, and will conduct human testing of the radioactive drug substance for safety and superiority compared to conventional iobenguane I 123 in normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* normal healthy volunteers with written informed consent who understand and are willing to comply with protocol requirements
* at least 21 years of age
* if female, then not of childbearing potential as documented by history (e.g., tubal ligation or hysterectomy) or is post menopausal with a minimum 1 year without menses
* if female of childbearing potential, a negative serum beta HCG pregnancy test within 24 hours prior to receiving iobenguane I 123
* if female of childbearing potential, agrees to use an acceptable form of birth control, defined as abstinence or use of IUD, oral contraceptive, barrier and spermicide, or hormonal implant, throughout the study period
* No existing predisposition to administration of thyroid blocking potassium iodide

Exclusion Criteria:

* females who are nursing
* documented history of significant allergy that required medical intervention to shellfish, X-ray contrast media, iodine/iodides, or iobenguane
* administered a radioisotope within 5 effective half-lives of that radioisotope prior to study enrollment
* abnormal screening laboratory studies (serum creatinine, SPOT, SGPT, total bilirubin as defined by standard laboratory reference ranges)
* those who have received an investigational compound and/or medical device within 30 days of entering this study
* pre-existing medical condition or circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study, (e.g. cancer, heart disease, or other medical conditions which potentially alter normal biodistribution)
* is determined by the investigator that the patient is clinically unsuitable for the study
* are taking medication which inhibits uptake of iobenguane I 123 within 2 weeks of enrollment, or tricyclic antidepressants or related drugs within 6 weeks of enrollment. Categories of medications include sympathomimetics, antihypertensives and cardiovascular agents, opioids, antipsychotics, tricyclic antidepressants, and medications as previously published
* have participated in a clinical trial with an investigational drug in the past 30 days.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Radiation dosimetry | 2 weeks
  Radiation dosimetry was measured by imaging at several time points. Blood and urine samples were also collected to correlate with imaging parameters. Side effects were also assessed after drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Bennett B Chin, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Chin BB, Kronauge JF, Femia FJ, Chen J, Maresca KP, Hillier S, Petry NA, James OG, Oldan JD, Armor T, Stubbs JB, Stabin MG, Babich JW. Phase-1 clinical trial results of high-specific-activity carrier-free 123I-iobenguane. J Nucl Med. 2014 May;55(5):765-71. doi: 10.2967/jnumed.113.124057. Epub 2014 Mar 13. PMID 24627436